CLINICAL TRIAL: NCT01594125
Title: An Open Label, Dose Escalation Phase I Study to Evaluate the Safety and Tolerability of Continuous Twice-daily Oral Treatment of Nintedanib in Japanese Patients With Hepatocellular Carcinoma.
Brief Title: Dose Escalation Study of Nintedanib (BIBF 1120) in Japanese Patients With Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1199.120
Record Dates: First submitted 2012-05-02; First posted 2012-05-08 (Estimated); Results first posted 2015-12-22 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-01

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — nintedanib

ARMS (2):
- Group I (Experimental): patients with mild liver dysfunction according to their AST/ALT values and Child-Pugh score
  Interventions: Drug: Nintedanib high dose; Drug: Nintedanib medium dose
- Group II (Experimental): patients with moderate liver dysfunction according to their AST/ALT values and Child-Pugh score
  Interventions: Drug: Nintedanib low dose; Drug: Nintedanib medium dose; Drug: Nintedanib high dose

INTERVENTIONS:
Drug: Nintedanib high dose — twice daily oral dosing
  Arms: Group I
Drug: Nintedanib low dose — twice daily oral dosing
  Arms: Group II
Drug: Nintedanib medium dose — twice daily oral dosing
  Arms: Group I
Drug: Nintedanib medium dose — twice daily oral dosing
  Arms: Group II
Drug: Nintedanib high dose — twice daily oral dosing
  Arms: Group II

SUMMARY:
The aim of the study is to investigate the safety, tolerability, efficacy and pharmacokinetics (PK) for Japanese hepatocellular carcinoma which are not amenable to curative surgery or loco regional therapy

ELIGIBILITY:
Inclusion criteria:

1. Histologically/cytologically confirmed hepatocellular carcinoma not amenable to curative surgery or loco-regional therapy
2. Age 20 years or older
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1
4. Child-Pugh score of 7 or less
5. Life expectancy more than 3 months
6. Time interval from last loco-regional therapy more than 4 weeks
7. Written informed consent in accordance with good clinical practice (GCP)

Exclusion criteria:

1. More than one line of prior systemic therapy for metastatic/unresectable hepatocellular carcinoma (HCC)
2. Fibrolamellar HCC
3. Uncontrolled or refractory ascites
4. Inadequate organ function
5. Variceal bleeding within 6 months or the presence of inappropriate varices
6. History of major thrombotic (except portal vein thrombosis) or clinically relevant major bleeding event in the past 6 months
7. Major surgery within 4 weeks
8. Known inherited predisposition to bleeding or thrombosis
9. Significant cardiovascular diseases

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-05; Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (5):
- Japan (5):
  - 1199.120.001 Boehringer Ingelheim Investigational Site, Chuo-ku, Tokyo
  - 1199.120.005 Boehringer Ingelheim Investigational Site, Fukuoka, Fukuoka
  - 1199.120.002 Boehringer Ingelheim Investigational Site, Kashiwa, Chiba
  - 1199.120.003 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1199.120.004 Boehringer Ingelheim Investigational Site, Saga, Saga

REFERENCES:
- [Derived] Okusaka T, Otsuka T, Ueno H, Mitsunaga S, Sugimoto R, Muro K, Saito I, Tadayasu Y, Inoue K, Loembe AB, Ikeda M. Phase I study of nintedanib in Japanese patients with advanced hepatocellular carcinoma and liver impairment. Cancer Sci. 2016 Dec;107(12):1791-1799. doi: 10.1111/cas.13077. Epub 2016 Dec 12. PMID 27627050

RESULTS

PARTICIPANT FLOW:
Groups:
- Group I: Nintedanib 150mg Bid: Patients with mild liver dysfunction according to their aspartate amino transferase (AST)/ alanine amino transferase (ALT) values (<=2 x upper limit of normal (ULN)) and Child-Pugh A treated with Nintedanib 150mg twice daily
- Group I: Nintedanib 200mg Bid: Patients with mild liver dysfunction according to their aspartate amino transferase (AST)/ alanine amino transferase (ALT) values (<=2 x upper limit of normal (ULN)) and Child-Pugh A treated with Nintedanib 200mg twice daily
- Group II: Nintedanib 100mg Bid: Patients with moderate liver dysfunction according to their aspartate amino transferase (AST)/ alanine amino transferase (ALT) values (>2 to <=5 x upper limit of normal (ULN)) and Child-Pugh B (score 7) treated with Nintedanib 100mg twice daily
- Group II: Nintedanib 150mg Bid: Patients with moderate liver dysfunction according to their aspartate amino transferase (AST)/ alanine amino transferase (ALT) values (>2 x to <=5 upper limit of normal (ULN)) and Child-Pugh B (score 7) treated with Nintedanib 150mg twice daily
- Group II: Nintedanib 200mg Bid: Patients with moderate liver dysfunction according to their aspartate amino transferase (AST)/ alanine amino transferase (ALT) values (>2 to <=5 x upper limit of normal (ULN)) and Child-Pugh B (score 7) treated with Nintedanib 200mg twice daily
Period: Overall Study
Arm/Group | Group I: Nintedanib 150mg Bid | Group I: Nintedanib 200mg Bid | Group II: Nintedanib 100mg Bid | Group II: Nintedanib 150mg Bid | Group II: Nintedanib 200mg Bid
Started | 4 | 12 | 3 | 4 | 7
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 12 | 3 | 4 | 7
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0
Not completed — Progressive Disease | 3 | 12 | 3 | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I: Nintedanib 150mg Bid | Group I: Nintedanib 200mg Bid | Group II: Nintedanib 100mg Bid | Group II: Nintedanib 150mg Bid | Group II: Nintedanib 200mg Bid | Total
Number analyzed (Participants) | 4 | 12 | 3 | 4 | 7 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (14.72) | 63.1 (9.84) | 73.3 (2.31) | 66.5 (6.56) | 67.4 (4.35) | 66.1 (8.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 2 | 1 | 9
  Male | 2 | 11 | 0 | 2 | 6 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities to Determine Maximum Tolerated Dose (MTD) of Nintedanib
Description: The MTD is based on the incidence of Dose Limiting Toxicities (DLTs). A drug-related AE was considered as a DLT if one of the following met: CTCAE grade 4 thrombocytopenia of any duration, CTCAE grade 4 neutropenia lasting for ≥8 days, CTCAE grade 4 febrile neutropenia of any duration, CTCAE grade 3 or 4 non-haematologic toxicity (with the following exception: Alopecia, Vomiting, nausea, or diarrhoea with no adequate supportive care, Transient electrolyte abnormality, which resolves spontaneously or can be corrected with appropriate treatment within 3 days, Liver toxicity), Liver enzyme toxicity of AST, ALT, alkaline phosphatase [ALP] elevation >5x ULN, or total bilirubin >3x ULN if baseline liver enzymes are within the normal range, or AST, ALT or ALP > baseline value + 4x ULN if the baseline value is elevated. The MTD was determined to be 200mg bid.
Time Frame: up to 28 days
Population: Patients from the MTD set: The MTD set contains only treated patients from the dose escalation that were not replaced for MTD determination.
Measure: Number; unit: participants
Arm/Group | Group I: Nintedanib 150mg Bid | Group I: Nintedanib 200mg Bid | Group II: Nintedanib 100mg Bid | Group II: Nintedanib 150mg Bid | Group II: Nintedanib 200mg Bid
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
participants | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Objective Tumour Response According to Response Evaluation Criteria in Solid Tumors (RECIST) 1.0
Description: Objective response (Complete response (CR) + Partial response (PR), regardless of confirmation) is derived from a patient's best objective response by RECIST. Best objective response is calculated based on the "overall" visit response from each assessment. Best objective response represents the best response a patient has had during their time in the study up until progression, last evaluable assessment in the absence of progression or the start of subsequent anti-cancer therapy. For patients whose progression event is death, best objective response will be calculated based on data up until the last evaluable RECIST assessment prior to death.
Time Frame: up to 28 months
Population: Treated Set (TS): The treated set includes all patients who were administered at least one dose of any study medication.
Measure: Number; unit: participants
Arm/Group | Group I: Nintedanib 150mg Bid | Group I: Nintedanib 200mg Bid | Group II: Nintedanib 100mg Bid | Group II: Nintedanib 150mg Bid | Group II: Nintedanib 200mg Bid
Number analyzed (Participants) | 4 | 12 | 3 | 4 | 7
participants | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the duration from start date of the study treatment to PD according to RECIST 1.0, or any death whichever occurs earlier.
Time Frame: up to 28 months
Population: Patients from TS
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Group I: Nintedanib 150mg Bid | Group I: Nintedanib 200mg Bid | Group II: Nintedanib 100mg Bid | Group II: Nintedanib 150mg Bid | Group II: Nintedanib 200mg Bid
Number analyzed (Participants) | 4 | 12 | 3 | 4 | 7
months | 6.05 [0.95 to 8.25] | 2.76 [1.74 to 5.42] | 7.26 [3.68 to 7.39] | 2.40 [1.48 to 6.88] | 2.76 [0.95 to 5.62]

4. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the duration from the start date of the study treatment to PD according to RECIST 1.0.
Time Frame: up to 28 months
Population: Patients from TS
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Group I: Nintedanib 150mg Bid | Group I: Nintedanib 200mg Bid | Group II: Nintedanib 100mg Bid | Group II: Nintedanib 150mg Bid | Group II: Nintedanib 200mg Bid
Number analyzed (Participants) | 4 | 12 | 3 | 4 | 7
months | 6.05 [0.95 to 8.25] | 2.76 [1.74 to 5.42] | 7.26 [3.68 to 7.39] | 2.40 [1.48 to 6.88] | 2.76 [0.95 to 5.62]

5. Secondary Outcome: Number of Participants With Response by Alpha Fetoprotein (AFP)
Description: Response by AFP is defined as 20% or more decline in AFP between the baseline value and the AFP value after three courses (12 weeks) of therapy. If patients only receive two courses of therapy the AFP value after two courses (8 weeks) will be used for the analysis.
Time Frame: up to 28 months
Population: Patients from TS and AFP evaluation (>20μg/L) at baseline and post-baseline AFP assessment after two or three courses.
Measure: Number; unit: participants
Arm/Group | Group I: Nintedanib 150mg Bid | Group I: Nintedanib 200mg Bid | Group II: Nintedanib 100mg Bid | Group II: Nintedanib 150mg Bid | Group II: Nintedanib 200mg Bid
Number analyzed (Participants) | 3 | 6 | 3 | 2 | 4
participants | 2 | 1 | 1 | 1 | 1

ADVERSE EVENTS:
Time Frame: up to 67 days
Arm/Group | Group I: Nintedanib 150mg Bid | Group I: Nintedanib 200mg Bid | Group II: Nintedanib 100mg Bid | Group II: Nintedanib 150mg Bid | Group II: Nintedanib 200mg Bid
Serious Adverse Events (participants affected / at risk) | 0/4 | 4/12 | 1/3 | 2/4 | 3/7
Other Adverse Events (participants affected / at risk) | 4/4 | 12/12 | 3/3 | 4/4 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group I: Nintedanib 150mg Bid (N=4) | Group I: Nintedanib 200mg Bid (N=12) | Group II: Nintedanib 100mg Bid (N=3) | Group II: Nintedanib 150mg Bid (N=4) | Group II: Nintedanib 200mg Bid (N=7)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 2 | 1
Tumour embolism (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group I: Nintedanib 150mg Bid (N=4) | Group I: Nintedanib 200mg Bid (N=12) | Group II: Nintedanib 100mg Bid (N=3) | Group II: Nintedanib 150mg Bid (N=4) | Group II: Nintedanib 200mg Bid (N=7)
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 3
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 7 | 1 | 1 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Loose tooth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 7 | 0 | 4 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 6 | 0 | 3 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 1 | 2 | 3 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 4 | 0 | 1 | 2
Oedema (General disorders) | 0 | 1 | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 1 | 1 | 1 | 1
Pyrexia (General disorders) | 1 | 1 | 0 | 1 | 2
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 2 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 2 | 1 | 1
Amylase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 3 | 2 | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 1 | 3 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 1 | 0 | 2
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 1 | 1
Haemoglobin decreased (Investigations) | 0 | 1 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 2 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 4 | 1 | 4 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 2 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Parosmia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Ketonuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 2 | 1 | 0 | 0 | 3
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 1 | 0 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.